CLINICAL TRIAL: NCT00384358
Title: A Phase 2, Multicenter, Single-Blind, Randomized, Stratified, Standard-Of-Care Controlled, Feasibility And Safety Study Of rhBMP-2/CPM As An Adjuvant Therapy For Fractures Of The Proximal Femur
Brief Title: Feasibility And Safety Study Of rhBMP-2/CPM For Hip Fractures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3100N7-211; B1921004
Record Dates: First submitted 2006-10-03; First posted 2006-10-06 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Fractures
Keywords: Fractures
MeSH Terms: conditions — Fractures, Bone | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): 1.0 mg/mL rhBMP-2/CPM + surgical fixation
  Interventions: Drug: rhBMP-2/CPM
- B (Experimental): 2.0 mg/mL rhBMP-2/CPM + surgical fixation
  Interventions: Drug: rhBMP-2/CPM
- C (Other): Control: Surgical fixation
  Interventions: Other: surgical intervention alone

INTERVENTIONS:
Drug: rhBMP-2/CPM — one time injection of 3-5 mL test article at time of internal fracture fixation
  Arms: A
Drug: rhBMP-2/CPM — one time injection of 3-5 mL test article at time of internal fracture fixation
  Arms: B
Other: surgical intervention alone — surgical internal fixation of fracture defines the standard of care group
  Arms: C

SUMMARY:
The primary objective of this study is to assess the safety of administering rhBMP-2/CPM as an adjuvant to internal fixation in subjects with fractures of the proximal femur.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 or older.
* Acute fracture of the proximal femur: displaced femoral neck fracture or unstable intertrochanteric femur fracture.
* Anatomic reduction (open or closed) and internal fixation within 48 hours following injury using any one of the following fixation constructs: 1) multiple parallel interfragmentary screws; 2) sliding hip screw and side plate fixation; or 3) cephalomedullary nail.

Exclusion Criteria:

* Concurrent fractures of the ipsilateral or contralateral lower extremity that would impede performance on functional assessments.
* Previous arthroplasty of contralateral (unaffected) hip.
* Planned procedure(s) to stimulate fracture healing after internal fixation of the fractured hip.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2006-12; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The safety outcome is the incidence of secondary fracture displacement among subjects treated with rhBMP-2/CPM compared to those receiving standard surgical treatment (internal fixation) alone. | upon completion 6 months of follow-up

SECONDARY OUTCOMES:
To establish a satisfactory method of administering rhBMP-2/CPM to implement in a phase 3 efficacy trial in this clinical indication. | 6 months follow-up
To estimate the success and failure rates associated with key fracture outcomes. | 6 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (30):
- United States (8):
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Pinellas Park, Florida
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, New Brunswick, New Jersey
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, Elmhurst, New York
- Australia (5):
  - Pfizer Investigational Site, Liverpool, New South Wales
  - Pfizer Investigational Site, Herston, Queensland
  - Pfizer Investigational Site, Adelaide, South Australia
  - Pfizer Investigational Site, Melbourne, Victoria
  - Pfizer Investigational Site, Parkville, Victoria
- Canada (4):
  - Pfizer Investigational Site, Ajax, Ontario
  - Pfizer Investigational Site, Chatham, Ontario
  - Pfizer Investigational Site, Scarborough Village, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
- Finland (2):
  - Pfizer Investigational Site, Oulu
  - Pfizer Investigational Site, Turku
- France (2):
  - Pfizer Investigational Site, Créteil
  - Pfizer Investigational Site, Marseille
- Germany (2):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Münster
- Hungary (2):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Debrecen
- Norway (2):
  - Pfizer Investigational Site, Bergen
  - Pfizer Investigational Site, Oslo
- Pfizer Investigational Site, Link?ping, Sweden
- United Kingdom (2):
  - Pfizer Investigational Site, Edinburgh
  - Pfizer Investigational Site, Norwich

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3100N7-211&StudyName=Feasibility%20And%20Safety%20Study%20Of%20rhBMP-2/CPM%20For%20Hip%20Fractures